CLINICAL TRIAL: NCT03962738
Title: RandoMized, DOuble-bliNd, PlacebO-coNtrolled Trial Of Lasmiditan in a Single Migraine Attack in Japanese Patients SuFfering From Migraine With or WithoUt Aura - the MONONOFU Study
Brief Title: A Study Lasmiditan (LY573144) in a Single Migraine Attack in Japanese Participants With Migraine
Acronym: MONONOFU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17012; H8H-JE-LAIH (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- 50 milligram (mg) Lasmiditan (Experimental): 50 mg Lasmiditan tablet plus two placebo tablets (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- 100 mg Lasmiditan (Experimental): 100 mg Lasmiditan tablet plus two placebo tablets (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- 200 mg Lasmiditan (Experimental): 200 mg Lasmiditan (two 100 mg tablets) plus one placebo tablet (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
  Interventions: Drug: Lasmiditan; Drug: Placebo
- Placebo (Placebo Comparator): Placebo tablets (to match 50 mg, 100 mg, 200 mg Lasmiditan dose tablets) administered once orally to treat a single migraine attack.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144
  Arms: 100 mg Lasmiditan; 200 mg Lasmiditan; 50 milligram (mg) Lasmiditan
Drug: Placebo — Administered orally

SUMMARY:
This study will assess the efficacy and safety of lasmiditan in the acute treatment of a migraine attack in Japanese adult participants with or without aura.

ELIGIBILITY:
Inclusion Criteria:

* Participants with migraine with or without aura fulfilling the International Classification of Headache Disorders (ICHD)-2.
* History of disabling migraine for at least 1 year.
* Migraine Disability Assessment Test (MIDAS) score ≥11.
* Migraine onset before the age of 50 years.
* History of 3-8 migraine attacks per month and <15 headache days per month during the past 3 months.

Exclusion Criteria:

* Known hypersensitivity to lasmiditan, or to any excipient of lasmiditan oral tablets.
* History or evidence of hemorrhagic stroke, epilepsy, or any other condition placing the patient at increased risk of seizures.
* History of recurrent dizziness and/or vertigo including benign paroxysmal positional vertigo, Meniere's disease, vestibular migraine, and other vestibular disorders.
* History of diabetes mellitus with complications (diabetic retinopathy, nephropathy, or neuropathy).
* History of orthostatic hypotension with syncope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- Japan (34):
  - Takanoko Hospital, Matsuyama, Ehime
  - Ikeda Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Jinnouchi Neurosurgery Clinic, Kasuga-shi, Fukuoka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Kohnan Hospital, Kobe, Hyōgo
  - Nishinomiya Municipal Central Hospital, Nishinomiya, Hyōgo
  - Yamaguchi Clinic, Nishinomiya-shi, Hyōgo
  - Fujitsu Clinic, Kawasaki, Kanagawa
  - Sendai Headache and Neurology Clinic, Sendai, Miyagi
  - Okayama City General Medical Center Okayama City Hospital, Okayama, Okayama-ken
  - Chibune General Hospital, Osaka, Osaka
  - Takase internal medicine clinic, Toyonaka-shi, Osaka
  - Osoegawa Neurology Clinic, Saga, Saga-ken
  - Saitama Medical University Hospital, Iruma-Gun, Saitama
  - Saitama Neuropsychiatric Institute, Saitama, Saitama
  - Saino Clinic, Tokorozawa, Saitama
  - Dokkyo Medical University Hospital, Shimotsuga-Gun, Tochigi
  - Niwa Family Clinic, Chofu-shi, Tokyo
  - Sanno Clinic Shinagawa, Minato-ku, Tokyo
  - USUDA CLINIC for internal medicine, Setagaya-ku, Tokyo
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Fukuuchi Pain Clinic, Shinjuku-ku, Tokyo
  - Sakura Clinic Internal Medicine Neurology, Toyama, Toyama
  - Nagaseki Headache Clinic, Kai-Shi, Yamanashi
  - Doi Clinic Internal Medicine Neurology, Hiroshima
  - Tanaka neurosurgical clinic, Kagoshima
  - Umenotsuji Clinic, Kochi
  - Kumamoto City Hospital, Kumamoto
  - Tatsuoka Neurology Clinic, Kyoto
  - Ishikawa Clinic, Kyoto
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - Tominaga Hospital, Osaka
  - Japanese Red Cross Shizuoka Hospital, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Kitamura S, Imai N, Tanji Y, Ozeki A, Komori M. Lasmiditan in Japanese Patients with Common Migraine Comorbidities or Concomitant Medications: A Post Hoc Safety and Efficacy Analysis from the MONONOFU Study. J Pain Res. 2023 May 25;16:1725-1738. doi: 10.2147/JPR.S399567. eCollection 2023. PMID 37255987
- [Derived] Matsumori Y, Komori M, Tanji Y, Ozeki A, Sakai F. Rapid Onset and Sustained Efficacy of Lasmiditan Among Japanese Patients with Migraine: Prespecified Analyses of a Randomized Controlled Trial. Neurol Ther. 2022 Dec;11(4):1721-1734. doi: 10.1007/s40120-022-00403-2. Epub 2022 Sep 22. PMID 36136232
- [Derived] MacGregor EA, Komori M, Krege JH, Baygani S, Vincent M, Pavlovic J, Igarashi H. Efficacy of lasmiditan for the acute treatment of perimenstrual migraine. Cephalalgia. 2022 Dec;42(14):1467-1475. doi: 10.1177/03331024221118929. Epub 2022 Aug 18. PMID 35979677
- [Derived] Doty EG, Hauck PM, Krege JH, Komori M, Hake AM, Dong Y, Lipton RB. The Association Between the Occurrence of Common Treatment-Emergent Adverse Events and Efficacy Outcomes After Lasmiditan Treatment of a Single Migraine Attack: Secondary Analyses from Four Pooled Randomized Clinical Trials. CNS Drugs. 2022 Jul;36(7):771-783. doi: 10.1007/s40263-022-00928-y. Epub 2022 Jul 2. PMID 35779194
- [Derived] Hashimoto Y, Komori M, Tanji Y, Ozeki A, Hirata K. Lasmiditan for single migraine attack in Japanese patients with cardiovascular risk factors: subgroup analysis of a phase 2 randomized placebo-controlled trial. Expert Opin Drug Saf. 2022 Dec;21(12):1495-1503. doi: 10.1080/14740338.2022.2078302. Epub 2022 Jun 24. PMID 35748397
- [Derived] Krege JH, Lipton RB, Baygani SK, Komori M, Ryan SM, Vincent M. Lasmiditan for Patients with Migraine and Contraindications to Triptans: A Post Hoc Analysis. Pain Ther. 2022 Jun;11(2):701-712. doi: 10.1007/s40122-022-00388-8. Epub 2022 Apr 26. PMID 35471625

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A participant who was randomized but did not treat with the study intervention was considered to have completed the study if they did not discontinue throughout the 8 weeks of treatment period and attended Visit 3 End of Study (EoS) or Early Discontinuation (EDC).
Groups:
- Placebo: Placebo tablets (to match 50 mg, 100 mg, 200 mg Lasmiditan dose tablets) administered orally once to treat a single migraine attack.
- 50 Milligrams (mg) Lasmiditan: 50 mg Lasmiditan tablet plus two placebo tablets (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
Period: Overall Study
Arm/Group | Placebo | 50 Milligrams (mg) Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Started | 258 | 109 | 261 | 218
Received At Least One Dose of Study Drug | 214 | 87 | 208 | 182
Completed | 251 | 109 | 259 | 217
Not Completed | 7 | 0 | 2 | 1
Not completed — Protocol Deviation | 3 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 50 mg Lasmiditan: 50 mg Lasmiditan tablet plus two placebo tablets (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
- Total: Total of all reporting groups
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan | Total
Number analyzed (Participants) | 214 | 87 | 208 | 182 | 691
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (8.95) | 44.9 (10.20) | 45.7 (9.66) | 44.7 (10.36) | 45.2 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 75 | 176 | 145 | 574
  Male | 36 | 12 | 32 | 37 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 214 | 87 | 208 | 182 | 691
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 214 | 87 | 208 | 182 | 691

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Headache Pain Free In High Dose Group (200 mg Lasmiditan)
Description: Percentage of participants who were headache pain free (defined as moderate or severe pain becoming none) at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: All randomized participants who received at least one dose of study drug to treat a migraine attack within 4 hours of onset and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 200 mg Lasmiditan
Number analyzed (Participants) | 211 | 179
percentage of participants | 16.6 | 40.8
Statistical Analysis 1: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.46, 95% CI 2-sided [2.17 to 5.54]

2. Secondary Outcome: Percentage of Participants Who Are Headache Pain Free in Each Dose Group
Description: Percentage of participants who are headache pain free in each dose group at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: All randomized participants who received one dose of study drug to treat a single migraine attack within 4 hours of onset and had postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 211 | 85 | 207 | 179
percentage of participants | 16.6 | 23.5 | 32.4 | 40.8
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan vs 100 mg Lasmiditan vs 200 mg Lasmiditan; Test type: Superiority; p < .001, Cochran-Armitage Trend Test

3. Secondary Outcome: Percentage of Participants With Headache Pain Relief
Description: Percentage of participants with headache pain relief (defined as moderate or severe headache pain becoming mild or none) at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Groups:
- 50 mg Lasmiditan: 50 mg Lasmiditan plus two placebo tablets (to match Lasmiditan dose) administered once orally to treat a single migraine attack.
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 211 | 85 | 207 | 179
percentage of participants | 55.0 | 68.2 | 80.2 | 78.2
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.03 to 2.99]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.34, 95% CI 2-sided [2.16 to 5.17]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.95, 95% CI 2-sided [1.89 to 4.62]

4. Secondary Outcome: Percentage of Participants Who Are Free of Most Bothersome Symptoms (MBS) Associated With Migraine
Description: Percentage of participants defined as the associated symptom present and identified as MBS (nausea, photophobia, or phonophobia) prior to dosing and being absent at 2 hours postdose.
  Missing value at a particular time point was considered as "nonresponder."
Time Frame: 2 Hours Postdose
Population: All randomized participants who received at least one dose of study drug to treat a single migraine attack within 4 hours of onset and had postdose headache severity or symptom assessments. Participants with no symptoms at pre-dose were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 157 | 59 | 150 | 121
percentage of participants | 46.5 | 55.9 | 58.0 | 60.3
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.197, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.81 to 2.72]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.044, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.01 to 2.50]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.08 to 2.83]

5. Secondary Outcome: Percentage of Participants With 24-Hour Sustained Pain Freedom
Description: Percentage of participants who are headache pain free at 2 hours postdose and 24 hours postdose with no rescue medication.
Time Frame: 24 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had any postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 212 | 87 | 208 | 180
percentage of participants | 10.4 | 14.9 | 20.2 | 23.2
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.268, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.73 to 3.17]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.26 to 3.82]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.50 to 4.61]

6. Secondary Outcome: Percentage of Participants With 48-Hour Sustained Pain Freedom
Description: Percentage of participants who are headache pain free at 2 hours postdose and 48 hours postdose with no rescue medication.
Time Frame: 48 Hours Postdose
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 212 | 87 | 208 | 180
percentage of participants | 12.3 | 14.9 | 19.7 | 21.1
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.535, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.61 to 2.58]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.036, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.04 to 3.03]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.018, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.12 to 3.33]

7. Secondary Outcome: Percentage of Participants That Are Free of Phonophobia
Description: Percentage of participants that are free of phonophobia at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: All randomized participants who received at least one dose of drug and had any postdose headache severity or symptom assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 208 | 86 | 203 | 171
percentage of participants | 83.7 | 89.5 | 87.2 | 86.5
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.199, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.76 to 3.65]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.305, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.77 to 2.32]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.426, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.71 to 2.24]

8. Secondary Outcome: Percentage of Participants That Are Free of Photophobia
Description: Percentage of participants that are free of photophobia at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had any postdose headache severity or symptom assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 208 | 86 | 203 | 171
percentage of participants | 69.2 | 77.9 | 76.8 | 77.8
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.135, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.87 to 2.82]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.080, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.95 to 2.30]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.061, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.98 to 2.49]

9. Secondary Outcome: Percentage of Participants That Are Free of Nausea
Description: Percentage of participants that are free of nausea at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo tablet (plus matching Lasmiditan placebo to maintain the blind) administered orally once to treat a single migraine attack.
- 50 mg Lasmiditan: 50 mg Lasmiditan tablet (plus two placebo tablets to maintain the blind) administered orally once to treat a single migraine attack.
- 100 mg Lasmiditan: 100 mg Lasmiditan tablet (plus two placebo tablets to maintain the blind) administered orally once to treat a single migraine attack.
- 200 mg Lasmiditan: 200 mg Lasmiditan (two 100 mg tablets) plus one placebo tablet (to maintain the blind) administered orally once to treat a single migraine attack.
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 208 | 86 | 203 | 171
percentage of participants | 78.8 | 83.7 | 82.3 | 79.5
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.342, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.71 to 2.67]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.377, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.76 to 2.04]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.862, Regression, Logistic; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.63 to 1.72]

10. Secondary Outcome: Percentage of Participants That Are Free of Vomiting
Description: Percentage of participants that are free of vomiting at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 208 | 86 | 203 | 171
percentage of participants | 99.0 | 97.7 | 99.5 | 100.0

11. Secondary Outcome: Percentage of Participants With Pain Freedom
Description: Percentage of participants with pain freedom.
Time Frame: 1 Hour Postdose
Population: All randomized participants who received one dose of study drug to treat a single migraine attack within 4 hours of onset and have postdose headache severity or symptom assessments.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 211 | 85 | 207 | 179
percentage of participants | 1.4 | 4.7 | 11.6 | 12.8
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.112, Regression, Logistic; Odds Ratio (OR) = 3.43, 95% CI 2-sided [0.75 to 15.65]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.05, 95% CI 2-sided [2.68 to 30.55]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.19, 95% CI 2-sided [3.01 to 34.55]

12. Secondary Outcome: Percentage of Participants With Headache Pain Relief
Description: Percentage of participants with headache pain relief at 1 hour postdose.
Time Frame: 1 Hour Postdose
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 211 | 85 | 207 | 179
percentage of participants | 41.2 | 35.3 | 58.5 | 59.8
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.343, Regression, Logistic; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.46 to 1.31]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.37 to 2.98]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.42 to 3.20]

13. Secondary Outcome: Percentage of Participants With Freedom From Most Bothersome Symptom (MBS)
Description: Percentage of participants defined as the associated symptom present and identified as MBS (nausea, photophobia, or phonophobia) prior to dosing and being absent at 1 hour postdose.
Time Frame: 1 Hour Postdose
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 157 | 59 | 150 | 121
percentage of participants | 28.7 | 32.2 | 42.0 | 33.1
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.605, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.62 to 2.26]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.015, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.12 to 2.90]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.432, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.74 to 2.05]

14. Secondary Outcome: Percentage of Participants With No Disability
Description: Disability will be measured by determining the level of interference with normal activities with 4 response options including: not at all (0); mild interference (1), marked interference (2); and need complete bed rest (3). No Disability timing is defined as the first time when severity becomes 0.
  Percentage of participants who are responders defined as score = 0 at 1 hours postdose.
Time Frame: 1 Hour Postdose
Population: All randomized participants who received one dose of study drug and had any postdose headache severity or symptom assessments. Participants with 0 severity at baseline are excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 209 | 81 | 199 | 173
percentage of participants | 8.1 | 13.6 | 10.6 | 12.1
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.166, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.79 to 3.96]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.396, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.68 to 2.62]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.181, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.81 to 3.11]

15. Secondary Outcome: Percentage of Participants With No Disability
Description: Disability will be measured by determining the level of interference with normal activities with 4 response options including not at all (0); mild interference (1), marked interference (2); and need complete bed rest (3). No Disability timing is defined as the first time when severity becomes 0.
  Percentage of participants who are responders defined as score = 0 at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had any postdose headache severity or symptom assessments. Participants with 0 severity at baseline are excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 206 | 85 | 201 | 171
percentage of participants | 18.4 | 24.7 | 25.4 | 28.7
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.233, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.79 to 2.64]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.092, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.94 to 2.41]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.017, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.11 to 2.92]

16. Secondary Outcome: Change From Baseline on the EuroQol 5 Dimension 5-level Scale (EQ-5D-5L) Health Status Index Score Japan
Description: The EQ-5D-5L was assessed based the EQ-5D-5L Health Status Index Score. The Japan specific tariffs (Japanese population-based index value) was used. The EQ-5D-5L is a participant rated, 2-part questionnaire. The first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that have 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The health state index score was calculated based on the responses to the 5 dimensions, providing a single value on a scale from less than 0 (where 0 is a health state equivalent to death; negative values are valued as worse than death) to 1 (perfect health), with higher scores indicating better health utility.
Time Frame: Baseline, 24 Hours Postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 186 | 75 | 176 | 150
score on a scale | 0.200 (0.218) | 0.192 (0.192) | 0.224 (0.198) | 0.186 (0.192)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.724, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.240, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.548, ANCOVA

17. Secondary Outcome: Change From Baseline on the EuroQol 5 Dimension 5-level Scale (EQ-5D-5L) Visual Analog Scale
Description: The EQ-5D-5L is a participant rated, 2-part questionnaire. The second part of the questionnaire consists of a visual analog scale on which the participant rates their perceived health state from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Time Frame: Baseline, 24 Hours Postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 186 | 75 | 176 | 150
score on a scale | 20.785 (26.094) | 19.640 (25.927) | 21.341 (26.920) | 19.320 (24.860)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.719, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p = 0.823, ANCOVA
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p = 0.612, ANCOVA

18. Secondary Outcome: Percentage of Participants With Very Much or Much Better as Measured by the Patient Global Impression of Change (PGI-C)
Description: The PGI-C is a one-item questionnaire that asks participants to provide their impression of change since taking the medicine. The PGI-C is measured using a 7-point Likert scale, with 1 = very much better, 2 = much better, 3 = a little better, 4 = no change, 5 = a little worse, 6 = much worse, and 7 = very much worse. Percentage of participants who are responders defined as having rated their impression of change as "very much better" or "much better" at 2 hours postdose.
Time Frame: 2 Hours Postdose
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 212 | 87 | 208 | 180
percentage of participants | 23.6 | 35.6 | 44.7 | 48.3
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Test type: Superiority; p = 0.037, Regression, Logistic; Odds Ratio (OR) = 1.78, 95% CI 2-sided [1.04 to 3.07]
Statistical Analysis 2: Comparison: Placebo vs 100 mg Lasmiditan; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.75 to 4.06]
Statistical Analysis 3: Comparison: Placebo vs 200 mg Lasmiditan; Test type: Superiority; p < .001, Regression, Logistic; Odds Ratio (OR) = 3.27, 95% CI 2-sided [2.11 to 5.06]

19. Secondary Outcome: Health-Related Quality of Life (HRQoL) Total Score as Measured by the 24-Hour Migraine Quality of Life Questionnaire (MQoLQ)
Description: The HRQoL is a 15-item, self-administered questionnaire. The items cover 5 domains (work functioning, social functioning, energy and vitality, feelings and concerns, and migraine symptoms). Each domain consists of 3 questions answered on a 7-point scale there 1 indicates maximum impairment and 7 indicating no impairment. A domain score is calculated by summing the responses to the 3 questions and the domain score ranges from 3 to 21, where a lower score indicates greater impairment, and a higher score indicates less impairment. The questionnaire will be administered 24 hours after the study drug.
Time Frame: 24 Hours Postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
Number analyzed (Participants) | 187 | 74 | 177 | 152
score on a scale
  Work Functioning | 12.594 (4.129) | 13.392 (3.930) | 13.034 (4.176) | 12.368 (4.197)
  Social Functioning | 13.235 (4.915) | 13.865 (4.336) | 13.429 (4.857) | 13.118 (4.803)
  Energy and Vitality | 12.652 (4.412) | 12.905 (4.224) | 12.723 (4.580) | 12.309 (4.277)
  Feelings and Concerns | 11.674 (4.145) | 11.622 (4.190) | 12.028 (4.181) | 12.099 (4.197)
  Migraine Symptoms | 14.070 (3.870) | 14.703 (3.877) | 14.949 (3.544) | 14.895 (3.754)
Statistical Analysis 1: Comparison: Placebo vs 50 mg Lasmiditan; Work Functioning; Test type: Superiority; p = 0.162, ANOVA
Statistical Analysis 2: Comparison: Placebo vs 50 mg Lasmiditan; Social Functioning; Test type: Superiority; p = 0.356, ANOVA
Statistical Analysis 3: Comparison: Placebo vs 50 mg Lasmiditan; Energy and Vitality; Test type: Superiority; p = 0.696, ANOVA
Statistical Analysis 4: Comparison: Placebo vs 50 mg Lasmiditan; Feelings and Concerns; Test type: Superiority; p = 0.914, ANOVA
Statistical Analysis 5: Comparison: Placebo vs 50 mg Lasmiditan; Migraine Symptoms; Test type: Superiority; p = 0.226, ANOVA
Statistical Analysis 6: Comparison: Placebo vs 100 mg Lasmiditan; Work Functioning; Test type: Superiority; p = 0.310, ANOVA
Statistical Analysis 7: Comparison: Placebo vs 100 mg Lasmiditan; Social Functioning; Test type: Superiority; p = 0.684, ANOVA
Statistical Analysis 8: Comparison: Placebo vs 100 mg Lasmiditan; Energy and Vitality; Test type: Superiority; p = 0.864, ANOVA
Statistical Analysis 9: Comparison: Placebo vs 100 mg Lasmiditan; Feelings and Concerns; Test type: Superiority; p = 0.412, ANOVA
Statistical Analysis 10: Comparison: Placebo vs 100 mg Lasmiditan; Migraine Symptoms; Test type: Superiority; p = 0.025, ANOVA
Statistical Analysis 11: Comparison: Placebo vs 200 mg Lasmiditan; Work Functioning; Test type: Superiority; p = 0.619, ANOVA
Statistical Analysis 12: Comparison: Placebo vs 200 mg Lasmiditan; Social Functioning; Test type: Superiority; p = 0.824, ANOVA
Statistical Analysis 13: Comparison: Placebo vs 200 mg Lasmiditan; Energy and Vitality; Test type: Superiority; p = 0.476, ANOVA
Statistical Analysis 14: Comparison: Placebo vs 200 mg Lasmiditan; Feelings and Concerns; Test type: Superiority; p = 0.352, ANOVA
Statistical Analysis 15: Comparison: Placebo vs 200 mg Lasmiditan; Migraine Symptoms; Test type: Superiority; p = 0.044, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: All randomized participants who received at least one dose of study drug regardless of whether they underwent any study assessments.
  Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 50 mg Lasmiditan | 100 mg Lasmiditan | 200 mg Lasmiditan
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/87 | 0/208 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/87 | 0/208 | 0/182
Other Adverse Events (participants affected / at risk) | 50/214 | 44/87 | 147/208 | 147/182
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=214) | 50 mg Lasmiditan (N=87) | 100 mg Lasmiditan (N=208) | 200 mg Lasmiditan (N=182)
Palpitations (Cardiac disorders) | 3 (3) | 4 (4) | 9 (10) | 4 (4)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 4 (4) | 5 (5) | 7 (7)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scintillating scotoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Xanthopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 7 (7) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 11 (11) | 16 (17)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 5 (6) | 2 (2)
Asthenia (General disorders) | 1 (1) | 5 (5) | 14 (14) | 18 (18)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Discomfort (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 5 (5) | 7 (8)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 7 (7) | 3 (3)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 3 (3) | 6 (6) | 23 (24) | 21 (22)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 11 (11) | 7 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 18 (18) | 79 (80) | 91 (93)
Dizziness postural (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 12 (12) | 24 (25)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 11 (11) | 7 (7) | 44 (45) | 41 (41)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dissociative disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (3) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/178 (1) | 0/75 (0) | 1/176 (1) | 1/145 (1)
Menstrual disorder (Reproductive system and breast disorders) | 0/178 (0) | 0/75 (0) | 0/176 (0) | 1/145 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0/178 (0) | 0/75 (0) | 1/176 (1) | 0/145 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03962738/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT03962738/SAP_001.pdf